CLINICAL TRIAL: NCT04682899
Title: Procalcitonin-guided Initiation of Antibiotics in AECOPD Inpatients: a Multicenter Randomized Controlled Trial
Brief Title: A Trial of Procalcitonin in Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Bin Cao, professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAP-China PCT-AECOPD
Record Dates: First submitted 2020-12-08; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-10

CONDITIONS: Procalcitonin; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCT-guided antibiotic therapy (PCT group) (Experimental): Participants in the PCT group will complete a PCT test within 2 hours after randomization and the results will be sent back to the clinician by laboratory through the internal network of the hospital. The prescribing clinician will use the results of the PCT to help guide their antibiotic prescription decision. The detailed recommendations are as follows: if PCT<0.1ng/ml，strongly discouraged；if PCT (0.1-0.25ng/ml) and no sputum purulence, discouraged; if PCT (0.1-0.25ng/ml) and sputum purulence, Recommended; PCT>0.25 ng/ml, Strongly recommended.
  Interventions: Drug: procalcitonin-guided antibiotic therapy
- Guideline-guided antibiotic therapy (guideline group) (Active Comparator): Participants in the guideline group will also need to complete a PCT test within 2 hours after randomization, however, the laboratory will save the results and do not sent back to the clinician. The clinician will make an antibiotic prescribing decision on the basis of the recommendations of GOLD guideline. The guideline recommend the following patients to receive antibiotic therapy. Patients with exacerbations of COPD who have three cardinal symptoms: increase in dyspnea, sputum volume, and sputum purulence; have two of the cardinal symptoms, if increased purulence of sputum is one of the two symptoms; or require mechanical ventilation (invasive or noninvasive).
  Interventions: Drug: guideline-guided antibiotic therapy

INTERVENTIONS:
Drug: procalcitonin-guided antibiotic therapy — In procalcitonin group, clinican make a decision of antibiotic precription based on the results of procalcitonin.
  Arms: PCT-guided antibiotic therapy (PCT group)
Drug: guideline-guided antibiotic therapy — In guideline group, clinican make a decision of antibiotic precription based on the recommendations of GOLD guideline.
  Arms: Guideline-guided antibiotic therapy (guideline group)

SUMMARY:
Current antibiotic prescription for patients with acute exacerbation of chronic obstructive pulmonary disease (AECOPD) is generally based on the Anthonisen criteria in The Global Initiative for Chronic Obstructive Pulmonary Disease (GOLD) guideline, that has a potential risk of antibiotics overuse. The dilemma is to identify patients who are most likely to benefit from antibiotics while avoiding unnecessary antibiotic use. Procalcitonin (PCT), a more sensitive and specific biomarker of bacterial infection than other conventional laboratory tests, has the potential to determine those patients in whom antibiotics would be beneficial. It is unclear whether PCT-guided antibiotic therapy is safe and effective for inpatients with AECOPD. The investigators aim to conduct a 2-arm, multicenter randomized controlled trial in China to determine whether PCT-guided antibiotic therapy will reduce the antibiotic prescription rate for AECOPD without negatively impacting the treatment success rate, compared with the GOLD guideline antibiotic recommendations.

DETAILED DESCRIPTION:
This trial will recruit 500 hopitalized patients with AECOPD. The eligible participants will be randomly assigned to either PCT group or guideline group.The investigators aim to compare the efficacy and safety between PCT-gudied antibiotic therapy and guideline-guided antibiotic recommendations. The primary hypothesis is that PCT-guided antibiotic therapy will reduce the antibiotic prescription rate for AECOPD without negatively impacting the treatment success rate, compared with the GOLD guideline antibiotic recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with AECOPD
* ≥40 years of age
* Able to understand and communicate to ensure the completion of the trial
* Voluntary participation and provide written informed consent

Exclusion Criteria:

* Fever, Axillary temperature≥38°C
* Pneumonia identified by X-Ray or CT of the chest
* Severe respiratory failure requiring admittance to ICU
* Concurrent infection at another site (e.g. urinary tract infection)
* Immunosuppression secondary to chemotherapy, AIDS or malignant tumor of blood system
* Comorbidities requiring corticosteroids (prednisone 30mg/d or equivalent more than 30 days )
* Invasive mechanical ventilation
* Patients with malignant tumors receiving chemotherapy or radiotherapy
* Pregnancy
* Participation in another clinical trial
* Previously enrollment into the study
* Refuse to attend

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Antibiotic prescription rate | within 30 days post randomization
  proportion of patients receiving antibiotics for AECOPD
Treatment success rate | day 30 post randomization
  Treatment success is defined as cure (a complete resolution of signs and symptoms associated with the exacerbation) or improvement (a resolution or reduction of the symptoms and signs associated with the exacerbation, without new symptoms or signs).

SECONDARY OUTCOMES:
Antibiotic prescription rate | day 1 post randomization
  the proportion of patients receiving antibiotics for AECOPD
Hospital antibiotic exposure | from randomization to hospital discharge, up to 30 days
  the number of days of antibiotic consumed for AECOPD and the proportion of patients receiving antibiotic for AECOPD between randomization and hospital discharge
Length of hospital stay | from randomization to hospital discharge, up to 30 days
  the number of days of hospitalization through study completion, an average of 30 days
Rate of subsequent exacerbation | within 30 days post randomization
  proportion of patients present with subsequent acute exacerbation after recovery
rate of hospital readmission | from the date of discharge to day 30 post randomization
  proportion of patients admit to hospital due to AECOPD after discharge
overall mortality | within 30 days post randomization
  death from all cause
ICU admission rate | within 30 days post randomization
  proportion of patients admit to ICU
Change in COPD assessment test | from the baseline of hospital admission to day 30 post randomization
  the difference between the baseline of hospital admission and day 30 post randomization
Change in modified Medical Research Council (mMRC) score | from the baseline of hospital admission to day 30 post randomization
  the difference between the baseline of hospital admission and day 30 post randomization

REFERENCES:
- [Derived] Huang L, Wang J, Gu X, Sheng W, Wang Y, Cao B. Procalcitonin-guided initiation of antibiotics in AECOPD inpatients: study protocol for a multicenter randomised controlled trial. BMJ Open. 2021 Aug 5;11(8):e049515. doi: 10.1136/bmjopen-2021-049515. PMID 34353802